CLINICAL TRIAL: NCT02296281
Title: Safety and Efficacy Study of Pirfenidone to Treat Grade 2 or Above Radiation-induced Lung Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: Shanghai Genomics, Inc. (Industry); GNI-EPS Pharmaceuticals, Inc. (GNI Group) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNI-F647-1401
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Radiation Pneumonitis
MeSH Terms: conditions — Radiation Pneumonitis | interventions — pirfenidone

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pirfenidone capsules to treat grade 2 or above radiation-induced lung injury patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old (include 18 and 70 years), male or female
2. The pathological diagnosis of lung cancer, with non-small cell lung cancer (NSCLC) staging IIIA or IIIB, and small cell lung cancer (SCLC) in council deadline
3. General condition assessment, ECOG score of 0-1
4. Enough heart, liver and kidney function, such as AST, ALT, LDH≤2 times ULN such as plasma total bilirubin, creatinine ≤1.5 times ULN; hematopoietic function enough, such as neutrophils ≥4.0 x109 / L, platelets ≥100 x109 / L
5. The expected survival at 6 months or more
6. Subject is able to eat solid food
7. The initial radical thoracic radiotherapy treatment
8. The clinical diagnosis of radiation-induced lung injury in Grade 2 or above
9. The duration of radiation-induced lung injury in less than 1 month
10. Signed informed consent

Exclusion Criteria:

1. Radiation-induced lung injury has entered the chronic phase
2. A history of chronic bronchitis, emphysema, or a history of cor pulmonale
3. Lung resection surgery
4. Cancer progression
5. Pulmonary infection
6. Associated with other serious diseases: such as occurred within 6 months of myocardial infarction, uncontrolled diabetes etc.
7. With active peptic ulcer
8. Pregnant women and patients with mental disease
9. Those who participate in clinical trials of other drugs within 3 months
10. Investigator judge does not apply to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Changes in radiation-induced lung injury classification | 36 Weeks